CLINICAL TRIAL: NCT06477640
Title: Home Rehabilitation Improves Cardiac Effort in Pulmonary Arterial Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: United Therapeutics (Industry); Mayo Clinic (Other); University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Lachant, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00009399
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension PAH
MeSH Terms: interventions — Exercise; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Intervention Group (Experimental)
  Interventions: Behavioral: Exercise
- Standard of Care (Placebo Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Exercise — The intervention group will receive daily activity messages sent through SMS text message or email.The messages will provide daily exercises with heart rate guidance.
  Arms: Exercise Intervention Group
Behavioral: Standard of Care — The control group will receive daily non-descript messages to help with blinding and to eliminate the confounding variable of daily contact. The messages will not include activity tasks and will include phrases such as "I hope you have a good day".
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate whether a home rehabilitation program for patients diagnosed with Pulmonary Arterial Hypertension (PAH) will decrease Cardiac Effort (number of heart beats used during 6-minute walk test/walk distance) and improve quality of life. Ultimately, this information could help improve the management of patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Follows at University of Rochester Medical Center Pulmonary Hypertension Clinic.
* Adult patients (>18 years old) with right heart catheterization confirmed pulmonary hypertension (PAH) on stable vasodilator dosing for at least 30 days. No planned titrations will occur during the 12-week study. If during the study, the treating physician feels it is necessary for safety reasons to adjust dosing, the subject will remain in their assigned group.
* Access to a smart phone or email to receive daily messages. If patients do not have access to either, we will offer a smartphone with cellular service for use during the study to receive daily messages.
* Clinically stable by the investigator (i.e., we will not enroll patients who endorse ongoing improvement or clinical worsening at enrollment).
* The treating investigator (Dr. Lachant or Dr. White) will review the clinical data of an eligible patient and establish them as safe to participate prior to approaching the patient for enrollment (i.e. not in decompensated heart failure or with recurrent pre-syncopal episodes prior to enrollment).

Exclusion Criteria:

* Pregnancy.
* Pulmonary Hypertension Groups 2-5.
* Resting tachycardia >120 beats/m during screening.
* Inability to walk.
* WHO Functional Class IV
* Lack of access to email or text messaging.
* Inability to follow daily instructions. including the two home 6-minute walk tests during the initial monitoring period. This is to show compliance with the protocol.
* Participating in a self-reported rehabilitation or exercise program.
* Oxygen therapy of more than 6 L/min at rest.
* Principal Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in cardiac effort | baseline to 3 months
  Cardiac effort is the number of heartbeats used during the a six minute walk test divided by walk distance

SECONDARY OUTCOMES:
Mean change in six minutes walk distance | baseline to 3 months
  The amount of distance walked in six minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No